CLINICAL TRIAL: NCT05754996
Title: Efficacy and Safety of Nifuroxazide in the Treatment of Hepatic Encephalopathy in Egyptian Patients With Liver Cirrhosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mennat Allah Saeid Emam, Teaching assistant, Future University in Egypt
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CL (3202)
Record Dates: First submitted 2023-02-23; First posted 2023-03-06 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Hepatic Encephalopathy
Keywords: Clinical Hepatic Encephalopathy Staging Scale; Hepatic encephalopathy; Nifuroxazide
MeSH Terms: conditions — Hepatic Encephalopathy | interventions — nifuroxazide; Lactulose; Rifaximin

STUDY DESIGN:
Intervention Model Description: This is a pilot, open-label, randomized controlled trial.
  The recruited patients will be randomly allocated in one of two groups:
  Group I (The study group): patients will receive oral nifuroxazide: 800 mg daily in 4 divided doses for maximum 7 days and lactulose 30 to 60 mL peroral (PO) three times daily (TID) according to bowel movement (to produce 2 to 3 semisoft stools per day) plus rifaximin 550 mg twice daily.
  Group II (The control group): patients will receive the standard treatment : lactulose 30 to 60 mL PO TID according to bowel movement (to produce 2 to 3 semisoft stools per day) plus rifaximin 550 mg twice daily..
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- lactulose plus Rifaximin plus nifuroxazide (Experimental): Nifuroxazide dosing : 800 mg daily in 4 divided doses for 7 days Lactulose dosing : 30 to 60 mL PO TID to produce 2 to 3 semisoft stools per day.
  Rifaximin: 550 mg twice daily
  Interventions: Drug: Nifuroxazide; Drug: Lactulose; Drug: Rifaximin 550Mg Tab
- Lactulose plus Rifaximin (Active Comparator): Lactulose dosing : 30 to 60 mL PO TID to produce 2 to 3 semisoft stools per day.
  Rifaximin: 550 mg twice daily
  Interventions: Drug: Lactulose; Drug: Rifaximin 550Mg Tab

INTERVENTIONS:
Drug: Nifuroxazide — Nifuroxazide dosing : 200 mg capsule four times daily
  Arms: lactulose plus Rifaximin plus nifuroxazide
Drug: Lactulose — Lactulose dosing: 30-60 mL PO TID with goal 2-3 semisoft stools
Drug: Rifaximin 550Mg Tab — Rifaximin 550 MG twice daily

SUMMARY:
This is a pilot study designed to evaluate the efficacy and safety of nifuroxazide in the treatment of hepatic encephalopathy in patients with grade II-III hepatic encephalopathy

DETAILED DESCRIPTION:
Hepatic Encephalopathy (HE) is a central nervous system dysfunction caused by liver insufficiency and/or portosystemic shunting, manifesting as a wide spectrum of neurological or psychiatric abnormalities characterized by alteration of cognitive and motor function.

The pathogenesis of hepatic encephalopathy is believed to be due to increased nitrogenous substances, primarily ammonia, in the blood. The treatment goal is to reduce nitrogen load from the GI tract and to improve central nervous system (CNS) status.

Treatment options include lactulose administered orally and non-absorbable antibiotics.

Lactulose is nonabsorbable disaccharides that is currently used as first line agents for the treatment of HE. Its action is thought to be due to Colonic metabolism of lactulose to lactic acid results in acidification of the gut lumen. This favors conversion of ammonium (NH4) to ammonia (NH3) and the passage of ammonia from tissues into the lumen. Gut acidification inhibits ammoniagenic coliform bacteria, leading to increased levels of nonammoniagenic lactobacilli. Lactulose also works as a cathartic, reducing colonic bacterial load.

Nifuroxazide is an oral broad-spectrum nitrofuran antibiotic that is commonly used as an intestinal anti-infective agent. It is active against the majority of intestinal bacteria: Gram-positive (Staphylococcus family) and Gram-negative (Enterobacteriaceae family: Escherichia, Citrobacter, Enterobacter, Klebsiella, Salmonella, Shigella, Yersinia) and is therefore expected to decrease ammonia production and to reverse the symptoms of HE.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from liver cirrhosis aging above 18 years who will be admitted to hospital with neuropsychiatric condition suggestive of hepatic encephalopathy (grade II or III) confirmed by their known previous hepatic disease by history, clinical examination and laboratory investigations in the form of hyperammonemia with Model for End-Stage Liver Disease (MELD) score ≤ 25 and patients are able to swallow.

Exclusion Criteria:

* Patients with neurological or communication problems.
* Degenerative central nervous system (CNS) disease.
* Any significant psychiatric illness.
* Patients with previous intake of nifuroxazide and rifaximin within the last month.
* Presence of underlying renal impairment (serum creatinine ≥ 2 mg/dL).
* Alcohol consumption within prior 4 weeks.
* Non-hepatic metabolic encephalopathy.
* Anemia with hemoglobin level < 7 g/dL.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2023-03-12 (Actual); Primary Completion 2025-07-29 (Actual); Study Completion 2025-07-29 (Actual)

PRIMARY OUTCOMES:
Number of patients achieving complete reversal of hepatic encephalopathy | 7 days
  Complete reversal is defined as the reversibility of HE from grade 2 or 3 to grade 0 or 1 according to West Haven criteria
The time for complete reversal of HE | 7 days
Evaluating the efficacy of nifuroxazide in improving mental status by calculating CHESS score | 7 days
  Evaluating the efficacy by measuring serum ammonia at baseline and at end of treatment and calculating (CHESS) score at baseline and at end of treatment.

SECONDARY OUTCOMES:
Length of hospital stay | 7 days
the rate of adverse events occurring during the treatment | Maximum 7 days
  Number of patients who experienced adverse events such as abdominal pain, vomiting, nausea, flatulence, anorexia, rash and headache.
Number of patients transferred to ICU | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Mennat Allah S. Emam, Principal Investigator — Cairo University
Locations (1):
- National Hepatology and Tropical Medicine Research Institute (NHTMRI), Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided